CLINICAL TRIAL: NCT04983706
Title: An Exploratory Study of Optimizing the Core Number and Location for MRI/Ultrasound Fusion Targeted Prostate Biopsy
Brief Title: Optimization of the Core Number and Location for Targeted Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IUNU-PC-110
Record Dates: First submitted 2021-07-01; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI/Ultrasound Fusion Saturation Biopsy (Experimental)
  Interventions: Procedure: MRI/Ultrasound Fusion Saturation Biopsy

INTERVENTIONS:
Procedure: MRI/Ultrasound Fusion Saturation Biopsy — MRI/Ultrasound fusion saturation biopsy: the core number and location are designed according to the lession condition.

SUMMARY:
This study aims to investigate the effect of core number and location optimization for targeted prostate biopsy on pathological accuracy.

DETAILED DESCRIPTION:
This is a single-center prospective study. The investigators perform MRI/US image fusion targeted saturation biopsy on prostate lesions with PI-RADS score 4, to investigate the effect of core number and location optimization for targeted prostate biopsy on pathological accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. Men more than 18 years old with clinical suspicion of prostate cancer;
2. Serum PSA ≤ 20 ng/ml within the previous 3 months;
3. No evidence of PSA increase by noncancerous factors, such as catheterization, bladder stones, or urinary tract infection including bacterial prostatitis;
4. mpMRI PI-RADS V2.1 score ≥4, diameter of ≤2.5 cm；
5. Able to provide written informed consent.

Exclusion Criteria:

1. Prior prostate biopsy or prostate surgery;
2. Prior treatment for prostate cancer;
3. Contraindication to MRI (e.g. claustrophobia, pacemaker);
4. Contraindication to prostate biopsy;
5. Men in whom artifact would reduce the quality of the MRI.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
The significant prostate cancer detection rate with different combinations of core number and location in the targeted saturated biopsy area | When histology results available, at an expected average of 3 days post-biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China